CLINICAL TRIAL: NCT01280084
Title: The Effect of Labour Analgesia on Babies' Movements After Birth: An Actigraphic Study
Brief Title: Labour Analgesia and Movement in Babies
Acronym: LAMB
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-02900
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Labour Analgesia and Neonate Activity
Keywords: neonate activity; labour analgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- No labour analgesia/nitrous oxide: Women who use no analgesia during labour or who only used nitrous oxide.
- Systemic opioids: Women who receive only systemic opioids for analgesia during, either intravenously or intramuscularly
- Intermediate dose epidural fentanyl: Women who receive a total epidural fentanyl dose less than 150 micrograms
- High dose epidural fentanyl: Women who receive a total epidural fentanyl dose more than 150 micrograms

SUMMARY:
This study aims to measure movements in babies after they are born using an actigraph, a wristwatch-sized device worn on the ankle, which works similarly to the device used by runners to count the number of steps they have taken. We aim to compare the movements of babies whose mothers have received different types of pain relief in labour.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the potential utility of actigraphy, a non-invasive means of measuring an individual's movements, in distinguishing the effects of different types of maternal labour analgesia on babies after birth.

The study hypothesizes that actigraphic data can be used to differentiate the effects on neonates of different forms of maternal intrapartum analgesia. In particular, we hypothesize that infants of mothers who receive intrapartum opioid analgesia will demonstrate fewer movements than infants of mothers who receive epidural analgesia or those who receive nothing.

Whilst it is well known that drugs administered to mothers during labour can affect their babies, means of assessing this effect are complex and unreliable. A more objective means of assessing babies after birth is required, and actigraphy may represent a useful technique. Actigraphy has been used on babies in other studies in a variety of settings, including comparing babies born by different delivery modes (i.e. vaginal versus cesarean delivery) and at different gestations (i.e. term versus preterm), although none of these studies have considered maternal analgesia received prior to delivery as a possible influence on babies' movements after birth. Other studies that have looked at sleep parameters in babies, particularly measures of activity, have shown association with later indices of psychomotor development.

The objective of the study is to compare actigraph-derived movement data from babies whose mothers have received any of the commonly used analgesic techniques for labour at BC Women's Hospital.

This is a prospective observational study. Women will be assessed for eligibility for the study on admission to the labour ward. As one of the inclusion criteria is vaginal birth, women considered eligible on admission may become ineligible depending on their mode fo delivery. Information will be available to all women in the assessment rooms and consent will be specifically sought after they deliver and are deemed eligible. We plan to recruit the babies of mothers who receive analgesia in one of four categories: no analgesia or nitrous oxide only; systemically administered opioid analgesia only; epidural analgesia with an intermediate total dose of fentanyl (<150mcg); epidural analgesia with a high total dose of fentanyl (>150mcg). We recognize that women may receive several or even all of the different modalities of labour analgesia in the course of their delivery. In this situation, we will calculate the total dose fo opioid received by all routes and convert this to fentanyl equivalents for the purposes of analysis. Neonates of women who agree to participate will be fitted with an actigraph that will remain in place (except for removal for bathing) for 24 hours, or until discharge from hospital. Actigraphs are small, light-weight, wrist-watch-sized monitors that weight 16 grams. The actigraphs will be placed on the neonates' ankle, as this position has been reported to cause less disturbance to them. Parents of participating neonates will also be instructed in the use fo a daily dairy that will allow correlation of actigraphic movement data with events such as bathing (when the actigraph will necessarily be removed) and other external sources of movements (e.g. being rocked, breastfeeding).

ELIGIBILITY:
Inclusion Criteria:

* Neonates born to healthy women with singleton pregnancies who deliver vaginally at term gestation (> 37 weeks)
* Mothers aged 19 years or older and understand written and oral English
* Neonates who are neurologically healthy

Exclusion Criteria:

* Cesarean delivery; patients booked for cesarean delivery presenting in labour
* Maternal opioid dependence
* Maternal sedative or psychotropic medications
* Maternal combined spinal epidural (CSE) analgesia in labour
* Forceps delivery; 4th degree perineal tears
* Birth weight greater than 4.5 kg
* Intrapartum fetal heart rate abnormalities requiring immediate delivery
* Neonates of mothers who receive epidural morphine for post-delivery analgesia
* Neonates requiring admission to NICU
* Neonates with obvious congenital anomalies

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women who have vaginal deliveries at BC Women's Hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Neonates' mobile and immobile time in 24 hours | Within the first 24 hours of life
Neonates' number of mobile and immobile bouts in 24 hours | Within the first 24 hours of life
Total activity score | Within the first 24 hours of life

SECONDARY OUTCOMES:
Neonates' total sleep time in 24 hours, night-time sleep in 24 hours and day-time sleep in 24 hours | Within the first 24 hours of life
Neonates' total number of sleep bouts | Within the first 24 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Kronitz, MD, FRCPC, Principal Investigator — Department of Anesthesia BC Women's Hospital
Locations (1):
- British Columbia Women's Hospital, Vancouver, British Columbia, Canada